CLINICAL TRIAL: NCT06578156
Title: Physiologic Effects of Nasal High Flow on Exercise Tolerance in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Physiologic Effects of Nasal High Flow on Exercise Tolerance in COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: American Thoracic Society (Other)
Responsible Party: Principal Investigator, Saramaria Afanador Castiblanco, Assistant Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20240476
Record Dates: First submitted 2024-08-28; First posted 2024-08-29 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nasal High Flow Cannula (Experimental): Nasal High Flow cannula at 70 liters per minute for 30 minutes. Given that this is a cross-over study, participants on this arm will be then crossed over to Nasal Low Flow Cannula at less than or equal to 4 liters per minute with supplemental oxygen for 30 minutes
  Interventions: Device: Nasal High Flow Cannula; Device: Nasal Low Flow Cannula
- Nasal Low Flow Cannula (Active Comparator): Low Flow Nasal Cannula at less than or equal to 4 liters per minute with supplemental oxygen at patient's baseline for 30 minutes. Given that this is a cross-over study, participants on this arm will be then crossed over to High Flow Cannula at 70 liters per minute for 30 minutes
  Interventions: Device: Nasal High Flow Cannula; Device: Nasal Low Flow Cannula

INTERVENTIONS:
Device: Nasal High Flow Cannula — High flow nasal cannula is a device that provides heated and humidified high flow gases. In-person. Depending on participant's availability, up to 6 times
Device: Nasal Low Flow Cannula — Low flow nasal cannula is a device that provides low flow gases. In-person. Depending on participant's availability, up to 6 times

SUMMARY:
This study aims to assess whether to describe the effects of the administration of nasal high flow (NHF) at 70 liters per minute (L/min) in a 6-Minute Walk Test (6-MWT) among Chronic Obstructive Pulmonary Disease (COPD) patients and to characterize the association between self-reported dyspnea with and without NHF at 70 L/min following a 6-MWT.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* Age 18 years or older
* Diagnosis of COPD
* Ability to ambulate without assistance
* Use of low-flow nasal cannula ≤ 4 L/min or no supplemental oxygen (O2) at all

Exclusion Criteria:

* Pregnancy
* Being on bedrest
* Inability to consent or cooperate with the study
* Using of > 4 L/min of supplemental O2 or requiring non-invasive ventilation during the daytime
* Hemodynamic instability (resting heart rate > 130/minute, systolic blood pressure of ≤ 90 mmHg or ≥ 180 mmHg)
* Metal implants in the thoracic regions (pacemakers, Automatic Implantable Cardioverter Defibrillator (AICD), plates, screws, rods, and disc replacements)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | 30 minutes
  The object of the test is to walk as far as possible for six minutes. The subject will walk at a normal pace around a marked course for six minutes. The distance walked in meters over 6 minutes will be measured.

SECONDARY OUTCOMES:
Breathing measured by the Borg dyspnea scale | 30 minutes
  This is a patient self-reported scale to rate the difficulty of breathing. The scale ranges from 0 to 10, where "0" indicated no difficulty breathing, and "10" indicates a maximal breathing difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Saramaria Afanador Castiblanco, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No